CLINICAL TRIAL: NCT04201483
Title: Real-time Ultrasound Imaging as Feedback for Deep Cervical Extensors Activation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1574447392087
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Neck Disorder
MeSH Terms: interventions — delta 24-sterol reductase

STUDY DESIGN:
Intervention Model Description: This will be a randomized clinical trial, with parallel groups and a blinded assessor performed in accordance with CONSORT guidelines. Participants will be randomized into two exercise groups: "DCE exercise without RUSI feedback (DCE)" and "DCE exercise with RUSI feedback (DCE+RUSI)". Randomization will be conducted using computer-generated random numbers (Epidat® version 3.1). Allocation concealment will be ensured using opaque and sealed envelopes
Who Masked: Outcomes Assessor
Masking Description: Ultrasound measurements will be performed by the rater responsible of performing ultrasound measurements who will be blinded to the assigned group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCE group (Active Comparator): DCE exercise without RUSI feedback
  Interventions: Other: DCE without RUSI feedback
- DCE + RUSI group (Experimental): DCE exercise with RUSI feedback
  Interventions: Other: DCE + RUSI feedback about performance

INTERVENTIONS:
Other: DCE without RUSI feedback — Participants assigned to this group will perform an exercise known to selectively activate the semispinalis cervicis muscle
  Arms: DCE group
Other: DCE + RUSI feedback about performance — Participants in this group will perform the same exercise as the DCE group to selectively activate the semispinalis cervicis muscle but receiving RUSI feedback about correct performance
  Arms: DCE + RUSI group

SUMMARY:
The aim of this study will be to determine the value of adding real-time ultrasound imaging (RUSI) as an external feedback tool for teaching the contraction of the deep cervical extensors (DCE) in healthy subjects. The potential benefit of RUSI to facilitate activation of the DCE during a specific motor task as well as the retention capacity of this motor task after a short period of training will be investigated

DETAILED DESCRIPTION:
Participants will be randomly allocated into two exercise groups: "DCE exercise without RUSI feedback (DCE)" and "DCE exercise with RUSI feedback (DCE+RUSI)".

Participants assigned to DCE will perform an exercise known to selectively activate the semispinalis cervicis muscles. By the other hand, participants in the DCE+RUSI group will perform the same exercise as the DCE group to selectively activate the semispinalis cervicis muscle but receiving RUSI feedback about correct performance. In both groups, a total of 10 sets of 10 repetitions will be performed with one minute of rest between each set.

Ultrasound measurement will be used to asses the antero-posterior dimension (thickness) of the DCE both at rest and during contraction at the level of C4 at baseline, immediately after the DCE exercise activation protocol and one-week follow-up in order to evaluate retention capacity.

All participants will be asked to not perform any other cervical motor control exercise or exercise using RUSI feedback until the last time point assessment will be finished.

All participants will be asked to avoid any exercises or treatments for neck pain between sessions.

All ultrasound images will be analysed off-line using Image J software. Thickness and percent thickness change will be measured. The percent thickness change will be calculated by using the following equation: thickness contracted - thickness rest / thickness rest.

ELIGIBILITY:
Inclusion Criteria:

* No actual neck pain
* Being able to understand Spanish language

Exclusion Criteria:

* Neck pain in the last 3 months
* Previous surgery in the neck region
* Neurological diseases or any other condition that may alter voluntary muscle contraction
* Previous experience with cervical motor control training exercises
* Previous experience using RUSI as an external feedback tool in any other body area

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-02-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Deep cervical extensors function at baseline | Baseline
  Ultrasound measurements will be used to asses the antero-posterior dimension (thickness) of the deep cervical extensors both at rest and during contraction at the level of C4
Change of the deep cervical extensors function from baseline to immediately after intervention | From baseline to immediately after intervention
  Ultrasound measurements will be used to asses the antero-posterior dimension (thickness) of the deep cervical extensors both at rest and during contraction at the level of C4
Change of the deep cervical extensors function from baseline to one week after intervention | From baseline to one week after intervention
  Ultrasound measurements will be used to asses the antero-posterior dimension (thickness) of the deep cervical extensors both at rest and during contraction at the level of C4

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy. University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code